CLINICAL TRIAL: NCT03256058
Title: The Effect of Different Applications of Tourniquet on Total Knee Arthroplasty
Brief Title: Tourniquet Application on Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2017-052
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-08

CONDITIONS: Tourniquets; Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinflation after early deflation (Active Comparator): The tourniquet would be inflated immediately before incision and deflated after the use of the cement, and 10 minutes later (after the hardening of the cement) , reinflate the tourniquet and deflate at the end of the operation.The total time of tourniquet inflation is controlled within 90 minutes.
  Interventions: Procedure: Reinflation after early deflation
- Control (Placebo Comparator): The tourniquet would be inflated immediately before incision and deflated at the end of the operation. The inflation of tourniquet should not last more than 90 minutes.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Reinflation after early deflation — the tourniquet would be inflated immediately before incision and deflated after the use of the cement , and 10 minutes later (after the hardening of the cement) , reinflate the tourniquet and deflate at the end of the operation. The total time of tourniquet inflation is controlled within 90 minutes.
  Arms: Reinflation after early deflation
Procedure: Control — The tourniquet would be inflated immediately before incision and deflated at the end of the operation. The inflation of tourniquet should not last more than 90 minutes.
  Arms: Control

SUMMARY:
This is a randomized controlled trial designed to research the effects of different tourniquet applications on postoperative pain in patients undergoing total knee arthroplasty, and to guide early postoperative recovery.

DETAILED DESCRIPTION:
Sixty participants undergoing unilateral TKA would be recruited in this study. On one side, the tourniquet would be inflated immediately before incision and deflated after the use of the cement , and 10 minutes later(after the hardening of the cement) , reinflate the tourniquet and deflate at the end of the operation. On the other side the tourniquet would be inflated immediately before incision and deflated at the end of the operation.The total time of tourniquet inflation is controlled within 90 minutes. The postoperative pain, limb swelling , the score of surgical field, blood pressure during the operation, blood loss, operating time, transfusion rate, deep vein thrombosis (DVT) incidence and clinical outcomes would be monitored for comparison.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anesthesiologists Grade 1-3 Patients
* Undergoing unilateral total knee arthroplasty under general anesthesia
* Should be treated with tourniquet

Exclusion Criteria:

* Tourniquet inflation time is less than 1h, greater than 1.5h
* Abnormal coagulation function
* BMI < 20kg/m2 or > 35kg/m2
* History of cerebral infarction
* History of Peripheral vascular disease
* Anemia (hemoglobin<90g/L)
* Systolic blood pressure (SBP) ≥ 170mmHg
* Pregnant blood glucose > 10mmol/L or HbA1c > 8.5% of diabetic patients
* History of chronic narcotic use
* Participate in other clinical trials at the same time
* Asked to withdraw from the trial

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours post surgery
  tested by Visual Analogue Scale

SECONDARY OUTCOMES:
The rate of postoperative limb swelling | 24 hours post surgery, 48 hours post surgery
  test the perimeter of the surgary limb at four fingers under the inguen,then Calculate the rate by formula (postoperative perimeter-preoperative perimeter)/preoperative perimeter
Endothelin-1 | one minute before tourniquet inflation, tourniquet inflation for an hour, one minute before tourniquet deflation, fifteen minutes after tourniquet deflation
  tested by ELISA
Nitric Oxide | one minute before tourniquet inflation, tourniquet inflation for an hour, one minute before tourniquet deflation, fifteen minutes after tourniquet deflation
  tested by ELISA
Lac | one minute before tourniquet inflation, tourniquet inflation for an hour, one minute before tourniquet deflation, fifteen minutes after tourniquet deflation
  blood gas analysis mmol/L
Hemoglobin | one minute before tourniquet inflation, tourniquet inflation for an hour, one minute before tourniquet deflation, fifteen minutes after tourniquet deflation
  blood gas analysis g/L
partial pressure of oxygen in artery | one minute before tourniquet inflation, tourniquet inflation for an hour, one minute before tourniquet deflation, fifteen minutes after tourniquet deflation
  blood gas analysis mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Guanglei Wang, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published

REFERENCES:
- [Result] Rama KR, Apsingi S, Poovali S, Jetti A. Timing of tourniquet release in knee arthroplasty. Meta-analysis of randomized, controlled trials. J Bone Joint Surg Am. 2007 Apr;89(4):699-705. doi: 10.2106/JBJS.F.00497. PMID 17403789
- [Result] Hernandez AJ, Almeida AM, Favaro E, Sguizzato GT. The influence of tourniquet use and operative time on the incidence of deep vein thrombosis in total knee arthroplasty. Clinics (Sao Paulo). 2012 Sep;67(9):1053-7. doi: 10.6061/clinics/2012(09)12. PMID 23018303
- [Result] Silver R, de la Garza J, Rang M, Koreska J. Limb swelling after release of a tourniquet. Clin Orthop Relat Res. 1986 May;(206):86-9. PMID 3708997
- [Result] Butt U, Ahmad R, Aspros D, Bannister GC. Factors affecting wound ooze in total knee replacement. Ann R Coll Surg Engl. 2011 Jan;93(1):54-6. doi: 10.1308/003588410X12771863937124. Epub 2010 Sep 10. PMID 20836920
- [Result] Palmer SH, Graham G. Tourniquet-induced rhabdomyolysis after total knee replacement. Ann R Coll Surg Engl. 1994 Nov;76(6):416-7. PMID 7702328
- [Result] Gielen MJ, Stienstra R. Tourniquet hypertension and its prevention: a review. Reg Anesth. 1991 Jul-Aug;16(4):191-4. No abstract available. PMID 1911493
- [Result] Kaufman RD, Walts LF. Tourniquet-induced hypertension. Br J Anaesth. 1982 Mar;54(3):333-6. doi: 10.1093/bja/54.3.333. PMID 6461346
- [Result] Valli H, Rosenberg PH. Effects of three anaesthesia methods on haemodynamic responses connected with the use of thigh tourniquet in orthopaedic patients. Acta Anaesthesiol Scand. 1985 Jan;29(1):142-7. doi: 10.1111/j.1399-6576.1985.tb02175.x. PMID 3976320
- [Result] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159
- [Result] Valli H, Rosenberg PH, Kytta J, Nurminen M. Arterial hypertension associated with the use of a tourniquet with either general or regional anaesthesia. Acta Anaesthesiol Scand. 1987 May;31(4):279-83. doi: 10.1111/j.1399-6576.1987.tb02566.x. PMID 3591250
- [Result] Bostankolu E, Ayoglu H, Yurtlu S, Okyay RD, Erdogan G, Deniz Y, Hanci V, Can M, Turan IO. Dexmedetomidine did not reduce the effects of tourniquet-induced ischemia-reperfusion injury during general anesthesia. Kaohsiung J Med Sci. 2013 Feb;29(2):75-81. doi: 10.1016/j.kjms.2012.08.013. Epub 2012 Oct 13. PMID 23347808
- [Result] Lin L, Wang L, Bai Y, Zheng L, Zhao X, Xiong X, Jin L, Ji W, Wang W. Pulmonary gas exchange impairment following tourniquet deflation: a prospective, single-blind clinical trial. Orthopedics. 2010 Jun 9;33(6):395. doi: 10.3928/01477447-20100429-15. PMID 20806768
- [Result] Matziolis G, Drahn T, Schroder JH, Krocker D, Tuischer J, Perka C. Endothelin-1 is secreted after total knee arthroplasty regardless of the use of a tourniquet. J Orthop Res. 2005 Mar;23(2):392-6. doi: 10.1016/j.orthres.2004.08.021. PMID 15734253
- [Result] Wang BQ, Kan YF, Yang QH. [The protective effect of the limb ischemia preconditioning on the hepatic injury related to NO/ET-1 system in rats]. Zhongguo Ying Yong Sheng Li Xue Za Zhi. 2010 Aug;26(3):376-9. Chinese. PMID 21038696
- [Result] Shao D, Park JE, Wort SJ. The role of endothelin-1 in the pathogenesis of pulmonary arterial hypertension. Pharmacol Res. 2011 Jun;63(6):504-11. doi: 10.1016/j.phrs.2011.03.003. Epub 2011 Mar 16. PMID 21419223
- [Result] Luscher TF, Barton M. Endothelins and endothelin receptor antagonists: therapeutic considerations for a novel class of cardiovascular drugs. Circulation. 2000 Nov 7;102(19):2434-40. doi: 10.1161/01.cir.102.19.2434. PMID 11067800
- [Result] Tarwala R, Dorr LD, Gilbert PK, Wan Z, Long WT. Tourniquet use during cementation only during total knee arthroplasty: a randomized trial. Clin Orthop Relat Res. 2014 Jan;472(1):169-74. doi: 10.1007/s11999-013-3124-2. PMID 23836239
- [Result] Mittal R, Ko V, Adie S, Naylor J, Dave J, Dave C, Harris IA, Hackett D, Ngo D, Dietsch S. Tourniquet application only during cement fixation in total knee arthroplasty: a double-blind, randomized controlled trial. ANZ J Surg. 2012 Jun;82(6):428-33. doi: 10.1111/j.1445-2197.2012.06083.x. Epub 2012 May 10. PMID 22571508
- [Result] Chen S, Li J, Peng H, Zhou J, Fang H, Zheng H. The influence of a half-course tourniquet strategy on peri-operative blood loss and early functional recovery in primary total knee arthroplasty. Int Orthop. 2014 Feb;38(2):355-9. doi: 10.1007/s00264-013-2177-x. Epub 2013 Nov 21. PMID 24258152
- [Result] Hernandez-Castanos DM, Ponce VV, Gil F. Release of ischaemia prior to wound closure in total knee arthroplasty: a better method? Int Orthop. 2008 Oct;32(5):635-8. doi: 10.1007/s00264-007-0376-z. Epub 2007 May 15. PMID 17503044
- [Result] Wauke K, Nagashima M, Kato N, Ogawa R, Yoshino S. Comparative study between thromboembolism and total knee arthroplasty with or without tourniquet in rheumatoid arthritis patients. Arch Orthop Trauma Surg. 2002 Nov;122(8):442-6. doi: 10.1007/s00402-002-0404-9. Epub 2002 Apr 18. PMID 12442180
- [Result] Sapega AA, Heppenstall RB, Chance B, Park YS, Sokolow D. Optimizing tourniquet application and release times in extremity surgery. A biochemical and ultrastructural study. J Bone Joint Surg Am. 1985 Feb;67(2):303-14. PMID 3968122
- [Result] Kadoi Y, Ide M, Saito S, Shiga T, Ishizaki K, Goto F. Hyperventilation after tourniquet deflation prevents an increase in cerebral blood flow velocity. Can J Anaesth. 1999 Mar;46(3):259-64. doi: 10.1007/BF03012606. PMID 10210051
- [Result] Huang CH, Wang MJ, Chen TL, Huang HH, Hsu HW, Susetio L, Liu CC. Blood and central venous pressure responses after serial tourniquet deflation during bilateral total knee replacement. J Formos Med Assoc. 1996 Jun;95(6):496-9. PMID 8772061